CLINICAL TRIAL: NCT02237482
Title: Is the Trabecular Metal Cup Associated With Lower Risk of Aseptic Loosening in Acetabular Revision Surgery?
Brief Title: Investigating Proximal Migration in Trabecular Metal Cups Used In Acetabular Revision Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maziar Mohaddes Ardebili, M.D., Sahlgrenska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 539-06
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Prosthesis Loosening
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small periacetabular bone defects (Experimental): Patients with cup loosening and small periacetabular bone defects
  Interventions: Device: Trilogy cup; Device: Trabecular metal cup (TM)
- Large periacetabular bone defects (Experimental): Patients with cup loosening and large periacetabular bone defects
  Interventions: Device: Trabecular metal cup (TM); Device: ZCA cup

INTERVENTIONS:
Device: Trilogy cup
  Arms: Small periacetabular bone defects
Device: Trabecular metal cup (TM)
Device: ZCA cup
  Arms: Large periacetabular bone defects

SUMMARY:
This study is intended to compare the proximal migration of the tantalum design (TM) with a cemented cup used in conjunction with bone allografting in cases with major bone loss. A group of patients with good periacetabular bone stock are included to analyse the differences between the tantalum and titanium design regarding risk of loosening and differences in clinical outcome measures. Radiostereometry (RSA) is used to accurately measure migration and rotation of the revision cups.

DETAILED DESCRIPTION:
Acetabular component loosening is often associated with periacetabular bone loss. Different approaches are described to address the bone defects in acetabular revision surgery. Several authors have reported inferior results when uncemented Titanium alloys and older porous coated designs are used in acetabular revisions with significant bone loss. Cemented fixation of the revision cup with impaction bone grafting (BIG), introduced more than three decades ago has today a thorough documentation. The Tantalum designs, with inherent properties such as high volumetric porosity, low modulus of elasticity and high friction against the bone, have been suggested to improve the fixation of the acetabular component. Several authors have been reporting promising short- and medium-term results using the TM designs in acetabular revisions with large periacetabular bone defects. Proximal migration measured with radiostereometry (RSA) has been suggested to predict risk for late aseptic loosening in hip prosthesis surgery. This study was primarily to compare the proximal migration of the tantalum design with a cemented cup used in conjunction with bone allografting in cases with major bone loss. A group of patients with good periacetabular bone stock are included to analyse the differences between the tantalum and titanium design. RSA is used to accurately measure migration and rotation of the revision cups.

ELIGIBILITY:
Inclusion Criteria:

All patients with a loose acetabular component, undergoing revision

Exclusion Criteria:

Patient not able to understand the intention of the study

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proximal migration measured with RSA | 24 month postoperatively.
  All patients have been recruited (operated on) by end of December 2011. Our primary intention is to follow all patients a minimum of two years with RSA.

SECONDARY OUTCOMES:
Patient reported outcome measures | first two years postoperatively
  Harris Hip Score

OTHER OUTCOMES:
Re-revision due to aseptic loosening or radiographical loosening | minimum13 years postoperative
EuroQol 5D | first two years postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Kärrholm, Professor, Study Director — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Borlin N, Rohrl SM, Bragdon CR. RSA wear measurements with or without markers in total hip arthroplasty. J Biomech. 2006;39(9):1641-50. doi: 10.1016/j.jbiomech.2005.05.004. Epub 2005 Jun 28. PMID 15990104
- [Background] Cuckler JM. Management strategies for acetabular defects in revision total hip arthroplasty. J Arthroplasty. 2002 Jun;17(4 Suppl 1):153-6. doi: 10.1054/arth.2002.32811. PMID 12068428
- [Background] Lakstein D, Backstein D, Safir O, Kosashvili Y, Gross AE. Trabecular Metal cups for acetabular defects with 50% or less host bone contact. Clin Orthop Relat Res. 2009 Sep;467(9):2318-24. doi: 10.1007/s11999-009-0772-3. Epub 2009 Mar 10. PMID 19277803
- [Background] Schreurs BW, Keurentjes JC, Gardeniers JW, Verdonschot N, Slooff TJ, Veth RP. Acetabular revision with impacted morsellised cancellous bone grafting and a cemented acetabular component: a 20- to 25-year follow-up. J Bone Joint Surg Br. 2009 Sep;91(9):1148-53. doi: 10.1302/0301-620X.91B9.21750. PMID 19721038